CLINICAL TRIAL: NCT02292693
Title: Comparison Three Different Laryngoscope Blades for Endotracheal Intubation in Pediatric Patients With Cervical Spine Immobilization.
Brief Title: Direct Laryngoscopy During Cervical Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/18
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Trauma
Keywords: intubation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intubation with immobilized cervical spine (Experimental): endotracheal intubation with immobilized cervical spine
  Interventions: Device: MIL; Device: MAC; Device: McCoy

INTERVENTIONS:
Device: MIL — Direct laryngoscopy. Laryngoscopy with Miller blade
Device: MAC — Direct laryngoscopy. Laryngoscopy with Macintosh blade
Device: McCoy — Direct laryngoscopy. Laryngoscopy with McCoy blade

SUMMARY:
The aim of this study was to compare time, success rates of different laryngoscope blades for intubation with an immobilized cervical spine in a standardized pediatric manikin model.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medicine personnel (physicians, nurses, paramedics)

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of first, second and third intubation attempts and overall effectiveness of intubation by participants

SECONDARY OUTCOMES:
Intubation time | 1 day
  time in seconds required for a successful intubation attempt
Cormack-Lehane grading | 1 day
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)
Preferred ETI device | 1day
  participants were asked which method of ETI they would prefer in a real-life resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland